CLINICAL TRIAL: NCT05490719
Title: A Single Arm, Phase II Clinical Study of Chemoradiationtherapy Combined With QL1706 (Anti-CTLA-4 and PD-1 Antibody) in Patients With Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Phase II Study of CRT Combined With QL1706 in ESCC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-IIT-02
Record Dates: First submitted 2022-07-11; First posted 2022-08-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Cancer; Concurrent chemoradiation; Immunotherapy; CTLA-4; PD-1; QL1706
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Radiation; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 plus Chemotherapy and Radiotherapy (Experimental): Radiotherapy: Total 50.4Gy/28 fraction ,1.8Gy per time，5 fractions per week.
  QL1706 will be administered at a dose of 5 mg/kg intravenously (IV), every 3 weeks, until progressive disease or intolerable or other reasons according to the criteria for termination of treatment). QL1706 will be administered up to 1 year.
  Chemotherapy: Taxol 135 mg/m2, days 1, 22; Cisplatin 25 mg/m2, day 1-3, day 22-24.
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — QL1706 is a humanized anti-PD1 IgG4 and anti-CTLA-4 IgG4 antibody.
  Other Names: Radiation; Taxol; Cisplatin

SUMMARY:
This is a single arm, multi-center Phase II Study. This clinical study is an investigator-initiated clinical trial（IIT). The objective of this study is to evaluate the efficacy and safety of Chemoradiationtherapy combined with QL1706 (anti-CTLA-4 and PD-1 antibody) in patients with unresectable locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participate voluntarily and sign informed consent.
2. age:18-75 years, male or female.
3. Histologically confirmed Advanced Unresectable Esophageal Squamous Cell Carcinomas,unresectable of clinical stage II-IVa patients (include unresectable,or surgical contraindication or refuse surgery)(According to AJCC 8th Edition stage , Pre-treatment clinical stage cT1N2-3M0,cT2-4bN0-3M0.
4. At least 1 measurable target lesion and/or unmeasurable target lesion according to Response Evaluation in Solid Tumors (RECIST 1.1).

Exclusion Criteria:

1. Patients who have a history of esophageal cancer surgery.
2. Previous history of fistula caused by primary tumor infiltration.
3. a high risk of gastrointestinal bleeding, esophageal fistula or esophageal perforation.
4. Subjects with poor nutritional status and weight loss of ≥ 10% in the first 2 months of screening have no significant improvement after nursing intervention.
5. Major surgery or serious trauma within 4 weeks before the first use of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by investigators | Up to approximately 2 years.
  Progression-free survival assessed by investigators

SECONDARY OUTCOMES:
OS | 1year and 3years
  Overall survival
ORR | Up to approximately 2 years
  Objective Response Rate，Complete Response plus Partial Response
DoR | Up to approximately 2 years
  Duration of Response
The rates and severity of Adverse Events, Serious Adverse Events | Through study completion, up to approximately 2 years
  The rates and severity of Adverse Events, Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin cancer hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhang W, Zhang T, Chen X, Li J, Gao L, Jiang S, Wang Y, Zheng Z, Dong J, Li Z, Zhao G, Cao F, Bai N, Wang P, Yan C, Pang Q. Iparomlimab and tuvonralimab (QL1706) combined definitive chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma (QL1706-IIT-02): a single arm, phase 2 trial. EClinicalMedicine. 2026 Jan 21;92:103758. doi: 10.1016/j.eclinm.2026.103758. eCollection 2026 Feb. PMID 41623855